CLINICAL TRIAL: NCT05087212
Title: A Single Arm, Open Label, Interventional Study Assessing the Mobilization Efficacy and Safety of Plerixafor in Combination With G- CSF in Multiple Myeloma Patients for Autologous Transplantation
Brief Title: Mobilization of Stem Cells With AMD3100 (Plerixafor) in Combination With G-CSF in Multiple Myeloma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16586; U1111-1266-4898 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-10-09; First posted 2021-10-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Autologous Haematopoietic Stem Cell Transplant
MeSH Terms: interventions — plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- plerixafor (Experimental): Participants will receive the first dose of plerixafor by subcutaneous (SC) injection on the evening of Day 4 (10 to 11 hours (± 1 hour) prior to the start of next day's apheresis). For a maximum of 4 days, patients will continue to receive daily plerixafor in the evening, followed by a morning dose of G-CSF and apheresis for up to a maximum of 4 apheresis or until ≥ 6×106 Cluster of differentiation 34 (CD34) + cells/kg were collected.
  Interventions: Drug: plerixafor + G-CSF

INTERVENTIONS:
Drug: plerixafor + G-CSF — subcutaneous (SC) injection

SUMMARY:
This is a single-group treatment, phase IV, open label study to assess the mobilization efficacy and safety of plerixafor in combination with G- CSF in male and female participants from 18 to 75 years of age with multiple myeloma for autologous transplantation. Study Duration-Screening-up to 30-day. Intervention and CD34+cells apheresis up-to 8 day. A follow up for 30 days (+7 days) post last dose of plerixafor, or the initiation of ablative chemotherapy, or the first dose of G-CSF administration in rescue procedure, whichever occurs earlier. Study duration up to 75 days. For treatment phase visit frequency-daily.

DETAILED DESCRIPTION:
The study duration consists of: An up-to 30-day screening, an up-to 8-day intervention and CD34+ cells apheresis and a follow up for 30 days (+7 days) post last dose of plerixafor, or the initiation of ablative chemotherapy, or the first dose of G-CSF administration in rescue procedure, whichever occurs earlier

ELIGIBILITY:
Inclusion Criteria:

* Participants must be with biopsy-confirmed diagnosis of multiple myeloma before the first mobilization, in first or second complete or partial remission
* The patient is eligible for autologous transplantation and treatment with an autologous peripheral Hematopoietic stem cell (HSC) transplant is planned
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Recovered from all acute toxic effects of prior chemotherapy or other cancer treatment
* Has an actual body weight <175% of their ideal body weight (IBW)
* In agreement to use an approved form of contraception if of childbearing potential

Exclusion Criteria:

* If they had a comorbid condition which, in the view of the investigators, rendered the patient at high risk from treatment complications
* Active brain metastases or myelomatous meningitis
* Abnormal Electrocardiogram (ECG) with clinically significant rhythm disturbance (ventricular arrhythmias), or other conduction abnormality in the last year that in the opinion of the investigator warrants exclusion of the subject from the trial.
* Active infection requiring antibiotic treatment
* Fever (temperature > 38°C)
* Positive pregnancy test in female patients
* Lactating females
* Had prior autologous or allogeneic transplantation
* Received bone-seeking radionuclides
* Received >6 cycles of induction therapy with lenalidomide
* Received >2 cycles of alkylating agent combinations
* Received more than 2 regimens of alkylating agent combinations
* Were less than 6 weeks off 1,3-bis(2-chloroethyl)-1- nitrosourea (BCNU) before first dose of G-CSF
* Were less than 4 weeks off last cycle of chemotherapy before first dose of G-CSF
* Failed previous hematopoietic stem cell collections or collection attempts
* Received radiation therapy to more than or equal to 50% of the pelvis
* Received specified treatment within specified duration.
* Patients whose apheresis product were to be further selected and purified
* Has received a live vaccine within 30 days of the planned start of study therapy. Seasonal flu vaccines that do not contain live virus are permitted
* Had previously received experimental therapy within 4 weeks of enrolling or currently enrolled in another experimental protocol
* White blood cell (WBC) count, Absolute neutrophil count (ANC)PLT count, estimated creatinine clearance, Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin should meet protocol requirements
* Positive test for HIV, active Hepatitis B (HBV), or active Hepatitis C (HCV) within 30 days prior to the first dose of IMP
* Has active central nervous system involvement
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or subjects who are legally institutionalized
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Participants are dependent on the Sponsor or Investigator
* Any specific situation during study implementation/course that may rise ethics considerations
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients collecting more than or equal to 6x106 CD34+ cells/kg in 2 or fewer apheresis days | Day 5 to Day 6

SECONDARY OUTCOMES:
the proportion of patients collecting more than or equal to 6x106 CD34+ cells/kg in 4 or fewer apheresis days | Day 5 to Day 8
the proportion of patients collecting more than or equal to 2x106 CD34+ cells/kg in 2 or fewer apheresis days | Day 5 to Day 6
the proportion of patients collecting more than or equal to 2x106 CD34+ cells/kg in 4 or fewer apheresis days | Day 5 to Day 8
the number of apheresis days required to reach more than or equal to 6x106 CD34+ cells/kg | Day 5 to Day 8
Peripheral Blood CD34+ count from Day 4 to Day 5 with the venous samples for Fluorescent activated cell sorting analysis obtained on the morning of Day 4 prior to administration of G-CSF and morning of Day 5 prior to administration of G-CSF | Day 4 to Day 5
Number of participants with Adverse events and Serious adverse events | Baseline to Day 30 (+7 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Sites, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16586 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25285&tenant=MT_SNY_9011